CLINICAL TRIAL: NCT01918826
Title: Evaluation of the Analgesic Efficiency of the Transcutaneous Neurostimulation in the Charcot Syndrome Marie Tooth on the Pains of Lower Limbs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-AOI-06
Record Dates: First submitted 2012-07-20; First posted 2013-08-08 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2012-07

CONDITIONS: CHARCOT MARIE TOOTH DISEASE
MeSH Terms: conditions — Charcot-Marie-Tooth Disease | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TENS active (Active Comparator): NEUROSTIMULATION TRANSCUTANEE AIMED ANALGESIC ACTIVE
  Interventions: Device: TENS
- TENS placebo (Placebo Comparator): NEUROSTIMULATION TRANSCUTANEE AIMED ANALGESIC PLACEBO
  Interventions: Device: TENS

INTERVENTIONS:
Device: TENS

SUMMARY:
The Charcot syndrome Marie Tooth is the most frequent hereditary neuromuscular diseases: there is no curative treatment at present, on the other hand precautionary measures can be taken (physiotherapy, port of splints, orthopaedic surgery and technical assistants). In the literature and in our recent study (evaluation of the pain in the disease of CMT - Reference center of the neuromuscular diseases - CHU Bow) the frequency of the pain is important varying from 66 to 96 % cases, affecting especially hands and lower limbs. The care of the pain in the Charcot syndrome Marie Tooth is not codified. The transcutaneous neurostimulation(TENS) is a not medicinal and not invasive therapeutics, without any brought back collateral effect, used at the same time in the chronic pain and acute since 1960, as well for the neuropathic pains that musculo-scrawny. No study was realized this day on the use of the TENS with analgesic aim in the CMT. We suggest studying the analgesic efficiency of the TENS in the Charcot syndrome Marie Tooth on the pains of lower limbs, the most frequent painful location in our recent works.

The main objective will be to analyze the improvement of the pain of lower limbs, based on the decrease of the analogical visual scale(ladder) (EVA), at least 30 %.

The secondary objectives will be to estimate repercussions on the functional capacities ( ONLS), the quality of life (SF(sci-fi) 12), the satisfaction (EVA), the global impression(printing) of change ( PGIC), the consumption of analgesic, DN4, NPSI (Neuropathic Pain Symptom Inventory), Concise Questionnaire of the Pains ( QCD), HAD (Hospital Anxiety and Depression scale).

ELIGIBILITY:
Inclusion Criteria:

* Age included between 18 and 75 years
* Affected by CMT confirmed on clinical, family criteria, electrophysiological and / or genetics
* pain ≥ 3 months
* EVA pain ≥ 4/10
* patient having given his written consent and lit(enlightened)
* patient susceptible to be followed regularly during at least 3 months
* Patient member to the Social Security

Exclusion Criteria:

* Expanding patients of associated neurological pathology
* Patients having resorted to the TENS in the last 3 months
* Medical history of cancers, collagen and quite other pathology which can interfere with the experimental procedure
* Patient carrier of a pacemaker or an active implantable medical device
* Cutaneous hurt on the territory to be stimulated
* Venous or arterial thrombosis or thrombophlebitis in the territory to be stimulated
* Patient participant in another biomedical research on the pain or the period of exclusion of which in a study is not ended
* Patient under guardianship or deprived of all his liberties

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | At 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Cécile RIBIERE, Principal Investigator — CHU NICE
Locations (1):
- CHU de Nice, Nice, France